CLINICAL TRIAL: NCT05366998
Title: Therapeutic Alliance and Treatment Outcome: A Study of the Private Clinic Hohenegg
Brief Title: Therapeutic Alliance and Treatment Outcome
Status: Completed | Type: Observational
Sponsor: Privatklinik Hohenegg (Other)
Responsible Party: Principal Investigator, Cosima Locher, Dr. phil., Privatklinik Hohenegg
Other Study IDs: 2021-01-070
Record Dates: First submitted 2022-04-28; First posted 2022-05-10 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Therapeutic Alliance
Keywords: Therapeutic Alliance; Treatment Outcome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to inform scientific understanding of the impact of the therapeutic alliance and the transition from inpatient to outpatient care.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to in-patient treatment in the private psychiatric clinic Hohenegg (PKH) from November 2021 onwards

Exclusion Criteria:

* Due to the naturalistic approach of the study, there will be no selection or exclusion made

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Patients who are admitted to the PKH. The PKH is a Swiss clinic with 70 beds, located in a rural setting. It treats patients in an inpatient setting for the following psychiatric disorders: depression, burnout, anxiety and psychosomatic disorders.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline psychological distress on Brief Symptom Checklist (BSCL, German version) at post-treatment and follow-up | Baseline, post-treatment (after 6-8 weeks) and follow-up (after 2-4 months)
  The BSCL is a 53-item self-report questionnaire that measures psychological distress and symptoms in the last seven days. Each item is rated on a 5-point Likert scale ranging from 0 = "not at all" to 4 = "extremely". The BSCL consists of nine different subscales: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism. Moreover, three global indices can be calculated: The Global Severity Index (GSI), providing information on psychological distress, the Positive Symptom Distress Index (PSDI), measuring the intensity of the reported symptoms, and the Positive Symptom Total (PST), indicating the number of present symptoms.

SECONDARY OUTCOMES:
Change from baseline quality of life on short version of the Incongruence Questionnaire (K-INK) at post-treatment and follow-up. | Baseline, post-treatment (after 6-8 weeks) and follow-up (after 2-4 months)
  The K-INK is a 23-item questionnaire and was developed as a short version of the INK with 93 items. It is based on the psychological construct of incongruence which is described as unsatisfactory realization of personal goals. These goals are based on the four basic psychological human needs, defined by Grawe, 1998 (Orientation and Control, Pleasure and Avoidance of pain, Self-Enhancement, Attachment). The items enquire information respective to these needs and are grouped in 14 respectively 9 scales: approach driven goals (one item per scale in the K-INK) and avoidance driven goals (one item per scale in the K-INK). Each item is rated on a 5-point Likert scale ranging from 0 = "(too) little" to 4 = "sufficient/satisfactory".
Change from baseline quality of life on the short version of the World Health Organization Quality of Life Instrument-Abbreviated Version (EUROHIS-QOL, German version) at post-treatment and follow-up | Baseline, post-treatment (after 6-8 weeks) and follow-up (after 2-4 months)
  The EUROHIS-QOL 8-Item Index is a short version of the WHOQOL-BREF containing 26 items grouped in four domains: physical, psychological, social relationships and environment. The EUROHIS-QOL 8-Item Index is composed of 2 items for each domain. The items are answered on a 5-point scale.
Change from post-treatment therapeutic alliance (inpatient treatment) on the short version of the Working Alliance Inventory - short revised (WAI-SR, German version) at follow-up (outpatient treatment) | Post-treatment (after 6-8 weeks) and follow-up (after 2-4 months)
  The WAI is a 12-item self-report questionnaire that measures the quality of alliance based on the following three aspects: the bond, the agreement on goals and the agreement on tasks. Each item is rated on a 5-point Likert scale ranging from 0 = "never" to 5 = "always". The WAI provides three subscales: bond, tasks and goals and one total scale.
Perceived social support in inpatient setting at post-treatment on the Fellow Patient Social Support (FEPB) | Post-treatment (after 6-8 weeks)
  The FEPB is a self-reported questionnaire and measures various aspects of the patient's social network during the clinical stay. In our study, we will use the 11th section, which assesses the overall impression of all relationships with fellow patients. The 11th section contains of eight items, whereby we will exclude item 4 and item 6 , because they do not fit the clinical.received by or due to fellow patients, each rated on a 5-point Likert scale ranging from 0 = "not at all" to 4 = "very much", as well as an item with an open question to qualitatively assess perceived support and distress from fellow patients. Moreover, the influence of fellow patients on treatment outcome is rated on a 5-point Likert scale from 0 = "very much worse" to 4 = "very much improved".
Perceived social support in outpatient setting at follow-up on the short version Social Support Questionnaire (F-SozU K-14, German Version) | follow-up (after 2-4 months)
  The F-SozU is a 14-item, self-reported questionnaire that measures perceived social support, whereby each item is rated on a 5-point Likert scale ranging from 1 = "not at all" to 5 = "completely". The questionnaire provides a global scale to assess the perceived social support based on emotional support, practical support and social integration.
Perceived helpfulness of therapy for therapist effect at post-treatment on a single item | Post-treatment (after 6-8 weeks)
  A single item, about the helpfulness of the different forms of therapy, rated on a 7-point Likert scale ranging from "not at all" to "extremely".
Perceived experience of loneliness at follow-up on the short version of the UCLA loneliness scale (UCLA, German version) | follow-up (after 2-4 months)
  The UCLA short version is a self-reported questionnaire that measures the feeling of loneliness with three items, each of which rated on a 3-point Likert scale ranging from 1 = "hardly ever" to 3 = "often". The UCLA yields a single scale, with higher scores indicating higher levels of loneliness.

OTHER OUTCOMES:
Perceived experience of the transition from the inpatient to the outpatient setting at post-treatment on a qualitative item | Post-treatment (after 6-8 weeks)
  A qualitative item about fears related to the transition to outpatient treatment.
Perceived experience of the transition from the inpatient to the outpatient setting at follow-up on qualitative items (Questions in this form are minimally adapted without changing intention due to the limited characters) | follow-up (after 2-4 months)
  14 qualitative items about
  * the transition to outpatient treatment
  * the influence of the PKH
  * maintaining contact to other patients
  * acquired skills from the inpatient treatment at PKH
  * improvements of the transition from inpatient to outpatient treatment
  * social support during the transition to outpatient treatment
Additional demographics; previous inpatient settings and significant events after the clinic at follow-up on qualitative items | follow-up (after 2-4 months)
  Two qualitative items, one about previous inpatient treatment experiences and the other about significant events after the treatment in the PKH.

CONTACTS AND LOCATIONS:
Overall Officials: Cosima A. Locher, Dr. phil., Principal Investigator — Privatklinik Hohenegg
Locations (1):
- Privatklinik Hohenegg, Meilen, Canton of Zurich, Switzerland